CLINICAL TRIAL: NCT05357963
Title: Incidence of Chronic Pain After Sternotomy
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Other Study IDs: E.Kurul-E1-22-2595
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain; Postoperative Pain, Acute; Postoperative Pain, Chronic; Sternotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sternotomy application — The chronic pain findings of the patients who underwent sternotomy will be questioned at the postoperative 3rd month.

SUMMARY:
Chronic postoperative pain is a well-known problem. Chronic postoperative pain is defined as pain that begins following a surgical procedure and persists for more than 2 months without other obvious causes such as infection or underlying disease. Sternotomy causes significant postoperative pain, and patients with chronic pain after sternotomy are often referred to pain clinics. The incidence of chronic pain after sternotomy ranges from 17% to 56%; In approximately one-third of these patients, chronic pain after sternotomy can compromise their quality of life by affecting their sleep patterns and impairing their ability to work. However, epidemiological studies on chronic pain after sternotomy are scarce. The aim of this study is to examine the incidence and possible risk factors of chronic pain following sternotomy operations. In this study, it was aimed to analyze the chronic pain findings of the patients who underwent sternotomy in the postoperative 3rd month.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists' physical status I-II-III-IV
* Body mass index (BMI) between 18-35 kg/m2
* Patients undergoing elective sternotomy

Exclusion Criteria:

* History of chronic analgesic therapy
* Patients with previous sternotomy surgery
* Patients who were operated under emergency conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-80 years, in the ASA I-II-III-IV risk group, with a BMI between 18-35 kg/m2 and undergoing sternotomy will be included in the study.
  Patients under the age of 18 years and over the age of 80 years, with an ASA score of V and above, with a BMI below 18 kg/m2 and above 35 kg/m2, who were operated under emergency conditions, and who received chronic pain treatment will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Chronic pain symptoms at 3rd months. | Chronic pain symptoms at 3rd month
  Chronic pain symptoms will be assessed using the numeric rating scale on a scale from 0 (no pain) to 10 (worst pain). Chronic pain symptoms (burning, stabbing, electric shock-like pain, tingling, numbness, pins, and needles feeling, hyperalgesia, allodynia, and hypoesthesia) will also be asked to the patients at the 3rd month after surgery.
Quality of life at 3rd months. | Quality of life at 3rd months.
  It will also be questioned whether the current pain of the patients affects their daily activities. It will be coded as '0 = not at all, 1 = slightly affecting, 2 = very affecting'.

SECONDARY OUTCOMES:
Acute pain score | At the 24th hour after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 24th hour after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün ZENGİN, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)